CLINICAL TRIAL: NCT00881595
Title: A Pilot Study Investigating Neoadjuvant Temozolomide-based Proton Chemoradiotherapy for High-Risk Soft Tissue Sarcomas
Brief Title: Proton Chemoradiotherapy for High-Risk Soft Tissue Sarcomas
Acronym: SA02
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No patients accrued since study opened
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UFPTI 0803-SA02
Record Dates: First submitted 2009-04-13; First posted 2009-04-15 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Soft Tissue Sarcomas
Keywords: Sarcomas; High-Risk Soft Tissue Sarcomas
MeSH Terms: conditions — Sarcoma | interventions — Temozolomide; Proton Therapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Proton Chemoradiotherapy followed by surgery (Other): Proton Chemoradiotherapy followed by surgery. Temozolomide five days per week during radiotherapy for 5 weeks. Proton radiation five days per week for 5 weeks Standard surgery will take place 4-6 weeks after completion of chemoradiation.
  Interventions: Procedure: Proton Chemoradiotherapy followed by surgery
- Chemoradiotherapy Temozolomide (Active Comparator): Chemoradiotherapy Temozolomide: 75 mg/m2 five days per week during radiotherapy for 5 weeks. Temozolomide should be taken orally 1 hour before each session of radiotherapy during weekdays (Monday through Friday). The dose will be determined using the body surface area (BSA) calculated at the beginning of the concurrent treatment. The BSA will be calculated from the height obtained at the pretreatment visit and the weight obtained before the first day of treatment. The concurrent treatment will last until the end of radiotherapy.
  Interventions: Drug: Chemoradiotherapy Temozolomide
- Proton Therapy (Active Comparator): 50 cobalt gray equivalent(CGE), 25 daily fractions, 5 weeks (2 CGE/fx)
  Interventions: Radiation: Proton therapy

INTERVENTIONS:
Drug: Chemoradiotherapy Temozolomide — Temozolomide: 75 mg/m2 five days per week during radiotherapy for 5 weeks.Temozolomide: 75 mg/m2 five days per week during radiotherapy for 5 weeks. Temozolomide should be taken orally 1 hour before each session of radiotherapy during weekdays (Monday through Friday). The dose will be determined using the body surface area (BSA) calculated at the beginning of the concurrent treatment. The BSA will be calculated from the height obtained at the pretreatment visit and the weight obtained before the first day of treatment. The concurrent treatment will last until the end of radiotherapy.
  Other Names: Temozolomide; Temodar
  Arms: Chemoradiotherapy Temozolomide
Radiation: Proton therapy — 50 cobalt gray equivalent(CGE), 25 daily fractions, 5 weeks (2 CGE/fx)
  Other Names: Radiation therapy
  Arms: Proton Therapy
Procedure: Proton Chemoradiotherapy followed by surgery — Proton Chemoradiotherapy followed by surgery. Resection of tumor at 4-6 weeks post-treatment.
  Arms: Proton Chemoradiotherapy followed by surgery

SUMMARY:
The goal of this study is to evaluate the effects of temozolomide and radiation combination in the treatment intended of soft tissue sarcomas.

This study will also look at the tumor tissue that was removed during your initial biopsy and your final surgery for information that may help to treat soft tissue sarcoma in the future. In addition the investigators will examine a sample of your normal tissue (optional) from the inside of your mouth/cheek (to compare it to your tumor tissue) before starting treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologic and radiographic proof of localized high-risk soft tissue sarcoma (STS) required prior to registration.
* For the purpose of this study, high risk STS is defined by at least two of the following risk factors:

  * Tumor ≥ 5 cm in maximal diameter on MRI or CT
  * Histology grade 3 or 4 (AJCC, 7th edition)
  * Tumor deep to the investing fascia
  * Locally recurrent sarcoma with no prior radiation therapy to the primary site
  * Age >55 years old
* Tumor must be considered potentially resectable as defined by cross sectional imaging.
* At least 2 weeks must have elapsed from any prior surgery or hormonal therapy. Patients must have ≤ grade 1 acute toxicities of any prior treatment with anti-cancer modalities (returned to baseline status as noted before most recent treatment). Patients with persisting, stable chronic toxicities from prior treatment ≤ grade 1 are eligible.
* Age ≥18 years at time of consent.
* Physician documented life expectancy of greater than 3 months.
* Patients must have normal organ and marrow function within 4 weeks prior to study treatment as defined below:

  * hemoglobin ≥ 9 g/dL
  * leukocytes ≥3,000/microliter (mcL)
  * absolute neutrophil count ≥1,500/mcL
  * platelets ≥100,000/mcL
  * total bilirubin ≤ institutional upper limit of normal
  * aspartate aminotransferase (AST/SGOT) and alanine aminotransferase(ALT/SGPT) < 2.5 x institutional upper limit of normal
  * creatinine within 1.5 x upper limit of normal(ULN)
* Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and for 12 months after treatment. Patients must have a negative serum pregnancy test within 14 days prior to beginning treatment on this trial. Sexually active men must also use appropriate contraception method and should not father a child while receiving therapy during this study.
* Ability to understand and the willingness to sign a written Institutional Review Board(IRB) stamped, study specific informed consent document prior to any research related procedures or study treatment.

Exclusion Criteria:

* Receiving any investigational agents.
* Treatment with cytotoxic agents and/or treatment with biologic agents within the 4 weeks prior to beginning treatment on this study.
* Evidence of metastatic disease.
* Previous radiotherapy to the affected site.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, and/or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because the investigational agents may have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with these agents, breastfeeding should be discontinued if the mother is treated.
* HIV-positive patients are ineligible because these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy and the potential pharmacokinetic interaction between antiretroviral therapy and the investigational agents.
* All herbal and/or alternative medications should be discontinued while on study, these include but are not limited to: Hydrastis canadensis (goldenseal), Uncaria tomentosa (cat's claw) or Echinacea angustifolia.
* Requirement for treatment with immunosuppressive agents or chronic steroids.
* A history of a hypersensitivity reaction to any of temozolomide's components or to Dacarbazine(DTIC).

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-02; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Assess treatment feasibility of neoadjuvant temozolomide-based proton chemoradiotherapy for high-risk soft tissue sarcoma | 6 months after surgery then every 6 months for 3 years

SECONDARY OUTCOMES:
Evaluate acute and late toxicities | Weekly during treatment, 6 months after surgery, then every 6 months for 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Indelicato, MD, Principal Investigator — University of Florida Proton Therapy Institute

REFERENCES:
- [Background] Anderson P, Aguilera D, Pearson M, Woo S. Outpatient chemotherapy plus radiotherapy in sarcomas: improving cancer control with radiosensitizing agents. Cancer Control. 2008 Jan;15(1):38-46. doi: 10.1177/107327480801500105. PMID 18094659
- [Background] Jemal A, Tiwari RC, Murray T, Ghafoor A, Samuels A, Ward E, Feuer EJ, Thun MJ; American Cancer Society. Cancer statistics, 2004. CA Cancer J Clin. 2004 Jan-Feb;54(1):8-29. doi: 10.3322/canjclin.54.1.8. PMID 14974761
- [Background] Pollock RE, Karnell LH, Menck HR, Winchester DP. The National Cancer Data Base report on soft tissue sarcoma. Cancer. 1996 Nov 15;78(10):2247-57. PMID 8918421
- [Background] Eilber FC, Rosen G, Nelson SD, Selch M, Dorey F, Eckardt J, Eilber FR. High-grade extremity soft tissue sarcomas: factors predictive of local recurrence and its effect on morbidity and mortality. Ann Surg. 2003 Feb;237(2):218-26. doi: 10.1097/01.SLA.0000048448.56448.70. PMID 12560780
- [Background] Pisters PW, Harrison LB, Leung DH, Woodruff JM, Casper ES, Brennan MF. Long-term results of a prospective randomized trial of adjuvant brachytherapy in soft tissue sarcoma. J Clin Oncol. 1996 Mar;14(3):859-68. doi: 10.1200/JCO.1996.14.3.859. PMID 8622034
- [Background] Rhomberg W, Hassenstein EO, Gefeller D. Radiotherapy vs. radiotherapy and razoxane in the treatment of soft tissue sarcomas: final results of a randomized study. Int J Radiat Oncol Biol Phys. 1996 Dec 1;36(5):1077-84. doi: 10.1016/s0360-3016(96)00433-6. PMID 8985029
- [Background] Rosenberg SA, Tepper J, Glatstein E, Costa J, Baker A, Brennan M, DeMoss EV, Seipp C, Sindelar WF, Sugarbaker P, Wesley R. The treatment of soft-tissue sarcomas of the extremities: prospective randomized evaluations of (1) limb-sparing surgery plus radiation therapy compared with amputation and (2) the role of adjuvant chemotherapy. Ann Surg. 1982 Sep;196(3):305-15. doi: 10.1097/00000658-198209000-00009. PMID 7114936
- [Background] Sindelar WF, Kinsella TJ, Chen PW, DeLaney TF, Tepper JE, Rosenberg SA, Glatstein E. Intraoperative radiotherapy in retroperitoneal sarcomas. Final results of a prospective, randomized, clinical trial. Arch Surg. 1993 Apr;128(4):402-10. doi: 10.1001/archsurg.1993.01420160040005. PMID 8457152
- [Background] Yang JC, Chang AE, Baker AR, Sindelar WF, Danforth DN, Topalian SL, DeLaney T, Glatstein E, Steinberg SM, Merino MJ, Rosenberg SA. Randomized prospective study of the benefit of adjuvant radiation therapy in the treatment of soft tissue sarcomas of the extremity. J Clin Oncol. 1998 Jan;16(1):197-203. doi: 10.1200/JCO.1998.16.1.197. PMID 9440743
- [Background] O'Sullivan B, Davis AM, Turcotte R, Bell R, Catton C, Chabot P, Wunder J, Kandel R, Goddard K, Sadura A, Pater J, Zee B. Preoperative versus postoperative radiotherapy in soft-tissue sarcoma of the limbs: a randomised trial. Lancet. 2002 Jun 29;359(9325):2235-41. doi: 10.1016/S0140-6736(02)09292-9. PMID 12103287
- [Background] Bonvalot S, Laplanche A, Lejeune F, Stoeckle E, Le Pechoux C, Vanel D, Terrier P, Lumbroso J, Ricard M, Antoni G, Cavalcanti A, Robert C, Lassau N, Blay JY, Le Cesne A. Limb salvage with isolated perfusion for soft tissue sarcoma: could less TNF-alpha be better? Ann Oncol. 2005 Jul;16(7):1061-8. doi: 10.1093/annonc/mdi229. Epub 2005 Jun 1. PMID 15930042
- [Background] Brennan MF. Staging of soft tissue sarcomas. Ann Surg Oncol. 1999 Jan-Feb;6(1):8-9. doi: 10.1007/s10434-999-0008-5. No abstract available. PMID 10030406
- [Background] Barkley HT Jr, Martin RG, Romsdahl MM, Lindberg R, Zagars GK. Treatment of soft tissue sarcomas by preoperative irradiation and conservative surgical resection. Int J Radiat Oncol Biol Phys. 1988 Apr;14(4):693-9. doi: 10.1016/0360-3016(88)90091-0. PMID 3350724
- [Background] Wunder JS, Nielsen TO, Maki RG, O'Sullivan B, Alman BA. Opportunities for improving the therapeutic ratio for patients with sarcoma. Lancet Oncol. 2007 Jun;8(6):513-24. doi: 10.1016/S1470-2045(07)70169-9. PMID 17540303
- [Background] Davis AM, O'Sullivan B, Turcotte R, Bell R, Catton C, Chabot P, Wunder J, Hammond A, Benk V, Kandel R, Goddard K, Freeman C, Sadura A, Zee B, Day A, Tu D, Pater J; Canadian Sarcoma Group; NCI Canada Clinical Trial Group Randomized Trial. Late radiation morbidity following randomization to preoperative versus postoperative radiotherapy in extremity soft tissue sarcoma. Radiother Oncol. 2005 Apr;75(1):48-53. doi: 10.1016/j.radonc.2004.12.020. PMID 15948265
- [Background] O'Sullivan B, Chung P, Euler C, Catton C. Soft Tissue Sarcoma. In: Gunderson LL, Tepper JE, editors. Clinical Radiation Oncology, ed. 2nd. Philadelphia: Elsevier; 2007:1519-1549.
- [Background] Bramwell V, Rouesse J, Steward W, Santoro A, Schraffordt-Koops H, Buesa J, Ruka W, Priario J, Wagener T, Burgers M, et al. Adjuvant CYVADIC chemotherapy for adult soft tissue sarcoma--reduced local recurrence but no improvement in survival: a study of the European Organization for Research and Treatment of Cancer Soft Tissue and Bone Sarcoma Group. J Clin Oncol. 1994 Jun;12(6):1137-49. doi: 10.1200/JCO.1994.12.6.1137. PMID 8201375
- [Background] Toma S, Canavese G, Grimaldi A, Ravera G, Ugolini D, Percivale P, Badellino F. Concomitant chemo-radiotherapy in the treatment of locally advanced and/or metastatic soft tissue sarcomas: experience of the National Cancer Institute of Genoa. Oncol Rep. 2003 May-Jun;10(3):641-7. PMID 12684637
- [Background] Cormier JN, Patel SR, Herzog CE, Ballo MT, Burgess MA, Feig BW, Hunt KK, Raney RB, Zagars GK, Benjamin RS, Pisters PW. Concurrent ifosfamide-based chemotherapy and irradiation. Analysis of treatment-related toxicity in 43 patients with sarcoma. Cancer. 2001 Sep 15;92(6):1550-5. doi: 10.1002/1097-0142(20010915)92:63.0.co;2-c. PMID 11745234
- [Background] Kraybill WG, Harris J, Spiro IJ, Ettinger DS, DeLaney TF, Blum RH, Lucas DR, Harmon DC, Letson GD, Eisenberg B; Radiation Therapy Oncology Group Trial 9514. Phase II study of neoadjuvant chemotherapy and radiation therapy in the management of high-risk, high-grade, soft tissue sarcomas of the extremities and body wall: Radiation Therapy Oncology Group Trial 9514. J Clin Oncol. 2006 Feb 1;24(4):619-25. doi: 10.1200/JCO.2005.02.5577. PMID 16446334
- [Background] Stevens MF, Hickman JA, Stone R, Gibson NW, Baig GU, Lunt E, Newton CG. Antitumor imidazotetrazines. 1. Synthesis and chemistry of 8-carbamoyl-3-(2-chloroethyl)imidazo[5,1-d]-1,2,3,5-tetrazin-4(3 H)-one , a novel broad-spectrum antitumor agent. J Med Chem. 1984 Feb;27(2):196-201. doi: 10.1021/jm00368a016. PMID 6694168
- [Background] Stevens MF, Hickman JA, Langdon SP, Chubb D, Vickers L, Stone R, Baig G, Goddard C, Gibson NW, Slack JA, et al. Antitumor activity and pharmacokinetics in mice of 8-carbamoyl-3-methyl-imidazo[5,1-d]-1,2,3,5-tetrazin-4(3H)-one (CCRG 81045; M & B 39831), a novel drug with potential as an alternative to dacarbazine. Cancer Res. 1987 Nov 15;47(22):5846-52. PMID 3664486
- [Background] Lunt E, Newton CG, Smith C, Stevens GP, Stevens MF, Straw CG, Walsh RJ, Warren PJ, Fizames C, Lavelle F, et al. Antitumor imidazotetrazines. 14. Synthesis and antitumor activity of 6- and 8-substituted imidazo[5,1-d]-1,2,3,5-tetrazinones and 8-substituted pyrazolo[5,1-d]-1,2,3,5-tetrazinones. J Med Chem. 1987 Feb;30(2):357-66. doi: 10.1021/jm00385a018. PMID 3806616
- [Background] Bull VL, Tisdale MJ. Antitumour imidazotetrazines--XVI. Macromolecular alkylation by 3-substituted imidazotetrazinones. Biochem Pharmacol. 1987 Oct 1;36(19):3215-20. doi: 10.1016/0006-2952(87)90636-8. PMID 2444229
- [Background] Tisdale MJ. Antitumour imidazotetrazines--XVIII. Modification of the level of 5-methylcytosine in DNA by 3-substituted imidazotetrazinones. Biochem Pharmacol. 1989 Apr 1;38(7):1097-101. doi: 10.1016/0006-2952(89)90254-2. PMID 2706009
- [Background] Tsang LL, Farmer PB, Gescher A, Slack JA. Characterisation of urinary metabolites of temozolomide in humans and mice and evaluation of their cytotoxicity. Cancer Chemother Pharmacol. 1990;26(6):429-36. doi: 10.1007/BF02994094. PMID 2225314
- [Background] Tsang LL, Quarterman CP, Gescher A, Slack JA. Comparison of the cytotoxicity in vitro of temozolomide and dacarbazine, prodrugs of 3-methyl-(triazen-1-yl)imidazole-4-carboxamide. Cancer Chemother Pharmacol. 1991;27(5):342-6. doi: 10.1007/BF00688855. PMID 1998993
- [Background] Buesa JM, Mouridsen HT, van Oosterom AT, Verweij J, Wagener T, Steward W, Poveda A, Vestlev PM, Thomas D, Sylvester R. High-dose DTIC in advanced soft-tissue sarcomas in the adult. A phase II study of the E.O.R.T.C. Soft Tissue and Bone Sarcoma Group. Ann Oncol. 1991 Apr;2(4):307-9. doi: 10.1093/oxfordjournals.annonc.a057942. PMID 1868027
- [Background] Gibson NW, Hickman JA, Erickson LC. DNA cross-linking and cytotoxicity in normal and transformed human cells treated in vitro with 8-carbamoyl-3-(2-chloroethyl)imidazo[5,1-d] -1,2,3,5-tetrazin-4(3H)-one. Cancer Res. 1984 May;44(5):1772-5. PMID 6713381
- [Background] Hartley JA, Gibson NW, Kohn KW, Mattes WB. DNA sequence selectivity of guanine-N7 alkylation by three antitumor chloroethylating agents. Cancer Res. 1986 Apr;46(4 Pt 2):1943-7. PMID 3004713
- [Background] Danson SJ, Middleton MR. Temozolomide: a novel oral alkylating agent. Expert Rev Anticancer Ther. 2001 Jun;1(1):13-9. doi: 10.1586/14737140.1.1.13. PMID 12113120
- [Background] Newlands ES, Blackledge GR, Slack JA, Rustin GJ, Smith DB, Stuart NS, Quarterman CP, Hoffman R, Stevens MF, Brampton MH, et al. Phase I trial of temozolomide (CCRG 81045: M&B 39831: NSC 362856). Br J Cancer. 1992 Feb;65(2):287-91. doi: 10.1038/bjc.1992.57. PMID 1739631
- [Background] Brada M, Judson I, Beale P, Moore S, Reidenberg P, Statkevich P, Dugan M, Batra V, Cutler D. Phase I dose-escalation and pharmacokinetic study of temozolomide (SCH 52365) for refractory or relapsing malignancies. Br J Cancer. 1999 Nov;81(6):1022-30. doi: 10.1038/sj.bjc.6690802. PMID 10576660
- [Background] Newlands ES, O'Reilly SM, Glaser MG, Bower M, Evans H, Brock C, Brampton MH, Colquhoun I, Lewis P, Rice-Edwards JM, Illingworth RD, Richards PG. The Charing Cross Hospital experience with temozolomide in patients with gliomas. Eur J Cancer. 1996 Dec;32A(13):2236-41. doi: 10.1016/s0959-8049(96)00258-4. PMID 9038604
- [Background] Bower M, Newlands ES, Bleehen NM, Brada M, Begent RJ, Calvert H, Colquhoun I, Lewis P, Brampton MH. Multicentre CRC phase II trial of temozolomide in recurrent or progressive high-grade glioma. Cancer Chemother Pharmacol. 1997;40(6):484-8. doi: 10.1007/s002800050691. PMID 9332462
- [Background] Reni M, Mason W, Zaja F, Perry J, Franceschi E, Bernardi D, Dell'Oro S, Stelitano C, Candela M, Abbadessa A, Pace A, Bordonaro R, Latte G, Villa E, Ferreri AJ. Salvage chemotherapy with temozolomide in primary CNS lymphomas: preliminary results of a phase II trial. Eur J Cancer. 2004 Jul;40(11):1682-8. doi: 10.1016/j.ejca.2004.03.008. PMID 15251157
- [Background] Garcia M, del Muro XG, Tres A, Crespo C, Valladares M, Lopez JJ, Rifa J, Perez X, Filipovich E, Germa-Lluch JR. Phase II multicentre study of temozolomide in combination with interferon alpha-2b in metastatic malignant melanoma. Melanoma Res. 2006 Aug;16(4):365-70. doi: 10.1097/01.cmr.0000215042.53683.40. PMID 16845333
- [Background] Lewis KD, Gibbs P, O'Day S, Richards J, Weber J, Anderson C, Zeng C, Baron A, Russ P, Gonzalez R. A phase II study of biochemotherapy for advanced melanoma incorporating temozolomide, decrescendo interleukin-2 and GM-CSF. Cancer Invest. 2005;23(4):303-8. doi: 10.1081/cnv-58832. PMID 16100942
- [Background] Brock CS, Newlands ES, Wedge SR, Bower M, Evans H, Colquhoun I, Roddie M, Glaser M, Brampton MH, Rustin GJ. Phase I trial of temozolomide using an extended continuous oral schedule. Cancer Res. 1998 Oct 1;58(19):4363-7. PMID 9766665
- [Background] Tolcher AW, Gerson SL, Denis L, Geyer C, Hammond LA, Patnaik A, Goetz AD, Schwartz G, Edwards T, Reyderman L, Statkevich P, Cutler DL, Rowinsky EK. Marked inactivation of O6-alkylguanine-DNA alkyltransferase activity with protracted temozolomide schedules. Br J Cancer. 2003 Apr 7;88(7):1004-11. doi: 10.1038/sj.bjc.6600827. PMID 12671695
- [Background] Spiro TP, Liu L, Majka S, Haaga J, Willson JK, Gerson SL. Temozolomide: the effect of once- and twice-a-day dosing on tumor tissue levels of the DNA repair protein O(6)-alkylguanine-DNA-alkyltransferase. Clin Cancer Res. 2001 Aug;7(8):2309-17. PMID 11489806
- [Background] Houghton PJ, Stewart CF, Cheshire PJ, Richmond LB, Kirstein MN, Poquette CA, Tan M, Friedman HS, Brent TP. Antitumor activity of temozolomide combined with irinotecan is partly independent of O6-methylguanine-DNA methyltransferase and mismatch repair phenotypes in xenograft models. Clin Cancer Res. 2000 Oct;6(10):4110-8. PMID 11051264
- [Background] Middlemas DS, Stewart CF, Kirstein MN, Poquette C, Friedman HS, Houghton PJ, Brent TP. Biochemical correlates of temozolomide sensitivity in pediatric solid tumor xenograft models. Clin Cancer Res. 2000 Mar;6(3):998-1007. PMID 10741727
- [Background] Aksoy S, Abali H, Kilickap S, Guler N. Successful treatment of a chemoresistant tumor with temozolomide in an adult patient: report of a recurrent intracranial mesenchymal chondrosarcoma. J Neurooncol. 2005 Feb;71(3):333-4. doi: 10.1007/s11060-004-1725-z. No abstract available. PMID 15735926
- [Background] Talbot SM, Keohan ML, Hesdorffer M, Orrico R, Bagiella E, Troxel AB, Taub RN. A phase II trial of temozolomide in patients with unresectable or metastatic soft tissue sarcoma. Cancer. 2003 Nov 1;98(9):1942-6. doi: 10.1002/cncr.11730. PMID 14584078
- [Background] Garcia del Muro X, Lopez-Pousa A, Martin J, Buesa JM, Martinez-Trufero J, Casado A, Poveda A, Cruz J, Bover I, Maurel J; Spanish Group for Research on Sarcomas. A phase II trial of temozolomide as a 6-week, continuous, oral schedule in patients with advanced soft tissue sarcoma: a study by the Spanish Group for Research on Sarcomas. Cancer. 2005 Oct 15;104(8):1706-12. doi: 10.1002/cncr.21384. PMID 16134177
- [Background] Stupp R, Mason WP, van den Bent MJ, Weller M, Fisher B, Taphoorn MJ, Belanger K, Brandes AA, Marosi C, Bogdahn U, Curschmann J, Janzer RC, Ludwin SK, Gorlia T, Allgeier A, Lacombe D, Cairncross JG, Eisenhauer E, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumor and Radiotherapy Groups; National Cancer Institute of Canada Clinical Trials Group. Radiotherapy plus concomitant and adjuvant temozolomide for glioblastoma. N Engl J Med. 2005 Mar 10;352(10):987-96. doi: 10.1056/NEJMoa043330. PMID 15758009
- [Background] Combs SE, Gutwein S, Schulz-Ertner D, van Kampen M, Thilmann C, Edler L, Wannenmacher MM, Debus J. Temozolomide combined with irradiation as postoperative treatment of primary glioblastoma multiforme. Phase I/II study. Strahlenther Onkol. 2005 Jun;181(6):372-7. doi: 10.1007/s00066-005-1359-x. PMID 15925979
- [Background] Chakravarti A, Erkkinen MG, Nestler U, Stupp R, Mehta M, Aldape K, Gilbert MR, Black PM, Loeffler JS. Temozolomide-mediated radiation enhancement in glioblastoma: a report on underlying mechanisms. Clin Cancer Res. 2006 Aug 1;12(15):4738-46. doi: 10.1158/1078-0432.CCR-06-0596. PMID 16899625
- [Background] Wedge SR, Porteous JK, Glaser MG, Marcus K, Newlands ES. In vitro evaluation of temozolomide combined with X-irradiation. Anticancer Drugs. 1997 Jan;8(1):92-7. doi: 10.1097/00001813-199701000-00013. PMID 9147618
- [Background] Lahiri DK, Song1 W, Ge YW. Analysis of the 5'-flanking region of the beta-amyloid precursor protein gene that contributes to increased promoter activity in differentiated neuronal cells. Brain Res Mol Brain Res. 2000 May 5;77(2):185-98. doi: 10.1016/s0169-328x(00)00051-6. PMID 10837914
- [Background] Raizer JJ, Malkin MG, Kleber M, Abrey LE. Phase 1 study of 28-day, low-dose temozolomide and BCNU in the treatment of malignant gliomas after radiation therapy. Neuro Oncol. 2004 Jul;6(3):247-52. doi: 10.1215/S1152851704000122. PMID 15279717
- [Background] Hegi ME, Diserens AC, Gorlia T, Hamou MF, de Tribolet N, Weller M, Kros JM, Hainfellner JA, Mason W, Mariani L, Bromberg JE, Hau P, Mirimanoff RO, Cairncross JG, Janzer RC, Stupp R. MGMT gene silencing and benefit from temozolomide in glioblastoma. N Engl J Med. 2005 Mar 10;352(10):997-1003. doi: 10.1056/NEJMoa043331. PMID 15758010
- [Background] Kawaguchi K, Oda Y, Saito T, Yamamoto H, Takahira T, Kobayashi C, Tamiya S, Tateishi N, Iwamoto Y, Tsuneyoshi M. DNA hypermethylation status of multiple genes in soft tissue sarcomas. Mod Pathol. 2006 Jan;19(1):106-14. doi: 10.1038/modpathol.3800502. PMID 16258501
- [Background] Temple CL, Ross DC, Magi E, DiFrancesco LM, Kurien E, Temple WJ. Preoperative chemoradiation and flap reconstruction provide high local control and low wound complication rates for patients undergoing limb salvage surgery for upper extremity tumors. J Surg Oncol. 2007 Feb 1;95(2):135-41. doi: 10.1002/jso.20629. PMID 17262730
- [Background] Virkus WW, Mollabashy A, Reith JD, Zlotecki RA, Berrey BH, Scarborough MT. Preoperative radiotherapy in the treatment of soft tissue sarcomas. Clin Orthop Relat Res. 2002 Apr;(397):177-89. doi: 10.1097/00003086-200204000-00022. PMID 11953609
- [Background] Nielsen OS, Cummings B, O'Sullivan B, Catton C, Bell RS, Fornasier VL. Preoperative and postoperative irradiation of soft tissue sarcomas: effect of radiation field size. Int J Radiat Oncol Biol Phys. 1991 Nov;21(6):1595-9. doi: 10.1016/0360-3016(91)90337-4. PMID 1938569
- [Background] Eilber FC, Eckardt JJ, Rosen G, Nelson SD, Selch M, Eilber FR. Large, deep, high-grade extremity sarcomas: treating tumors of the flexor fossae. Surg Oncol. 1999 Dec;8(4):211-4. doi: 10.1016/s0960-7404(00)00002-5. PMID 11128835
- [Background] Pollack A, Zagars GK, Goswitz MS, Pollock RA, Feig BW, Pisters PW. Preoperative vs. postoperative radiotherapy in the treatment of soft tissue sarcomas: a matter of presentation. Int J Radiat Oncol Biol Phys. 1998 Oct 1;42(3):563-72. doi: 10.1016/s0360-3016(98)00277-6. PMID 9806516
- [Background] Mack LA, Crowe PJ, Yang JL, Schachar NS, Morris DG, Kurien EC, Temple CL, Lindsay RL, Magi E, DeHaas WG, Temple WJ. Preoperative chemoradiotherapy (modified Eilber protocol) provides maximum local control and minimal morbidity in patients with soft tissue sarcoma. Ann Surg Oncol. 2005 Aug;12(8):646-53. doi: 10.1245/ASO.2005.03.064. Epub 2005 Jun 20. PMID 15965732
- [Background] Suit HD, Mankin HJ, Wood WC, Proppe KH. Preoperative, intraoperative, and postoperative radiation in the treatment of primary soft tissue sarcoma. Cancer. 1985 Jun 1;55(11):2659-67. doi: 10.1002/1097-0142(19850601)55:113.0.co;2-q. PMID 3995476
- [Background] Holt GE, Griffin AM, Pintilie M, Wunder JS, Catton C, O'Sullivan B, Bell RS. Fractures following radiotherapy and limb-salvage surgery for lower extremity soft-tissue sarcomas. A comparison of high-dose and low-dose radiotherapy. J Bone Joint Surg Am. 2005 Feb;87(2):315-9. doi: 10.2106/JBJS.C.01714. PMID 15687153
- [Background] Cannon CP, Ballo MT, Zagars GK, Mirza AN, Lin PP, Lewis VO, Yasko AW, Benjamin RS, Pisters PW. Complications of combined modality treatment of primary lower extremity soft-tissue sarcomas. Cancer. 2006 Nov 15;107(10):2455-61. doi: 10.1002/cncr.22298. PMID 17036354
- [Background] Goitein M, Jermann M. The relative costs of proton and X-ray radiation therapy. Clin Oncol (R Coll Radiol). 2003 Feb;15(1):S37-50. doi: 10.1053/clon.2002.0174. PMID 12602563
- [Background] Ogata T, Teshima T, Kagawa K, Hishikawa Y, Takahashi Y, Kawaguchi A, Suzumoto Y, Nojima K, Furusawa Y, Matsuura N. Particle irradiation suppresses metastatic potential of cancer cells. Cancer Res. 2005 Jan 1;65(1):113-20. PMID 15665286
- [Background] Paganetti H, Bortfeld T, Delaney TF. Neutron dose in proton radiation therapy: in regard to Eric J. Hall (Int J Radiat Oncol Biol Phys 2006;65:1-7). Int J Radiat Oncol Biol Phys. 2006 Dec 1;66(5):1594-5; author reply 1595. doi: 10.1016/j.ijrobp.2006.08.005. No abstract available. PMID 17126219
- [Background] Suit H, Kooy H, Trofimov A, Farr J, Munzenrider J, DeLaney T, Loeffler J, Clasie B, Safai S, Paganetti H. Should positive phase III clinical trial data be required before proton beam therapy is more widely adopted? No. Radiother Oncol. 2008 Feb;86(2):148-53. doi: 10.1016/j.radonc.2007.12.024. Epub 2008 Jan 30. PMID 18237800
- [Background] Griffin AM, Euler CI, Sharpe MB, Ferguson PC, Wunder JS, Bell RS, Chung PW, Catton CN, O'Sullivan B. Radiation planning comparison for superficial tissue avoidance in radiotherapy for soft tissue sarcoma of the lower extremity. Int J Radiat Oncol Biol Phys. 2007 Mar 1;67(3):847-56. doi: 10.1016/j.ijrobp.2006.09.048. Epub 2006 Dec 8. PMID 17161553
- [Background] Lin PP, Schupak KD, Boland PJ, Brennan MF, Healey JH. Pathologic femoral fracture after periosteal excision and radiation for the treatment of soft tissue sarcoma. Cancer. 1998 Jun 15;82(12):2356-65. PMID 9635528
- [Background] Tucker MA, D'Angio GJ, Boice JD Jr, Strong LC, Li FP, Stovall M, Stone BJ, Green DM, Lombardi F, Newton W, et al. Bone sarcomas linked to radiotherapy and chemotherapy in children. N Engl J Med. 1987 Sep 3;317(10):588-93. doi: 10.1056/NEJM198709033171002. PMID 3475572
- [Background] Hawkins MM, Wilson LM, Burton HS, Potok MH, Winter DL, Marsden HB, Stovall MA. Radiotherapy, alkylating agents, and risk of bone cancer after childhood cancer. J Natl Cancer Inst. 1996 Mar 6;88(5):270-8. doi: 10.1093/jnci/88.5.270. PMID 8614005
- [Background] Timmermann B, Schuck A, Niggli F, Weiss M, Lomax AJ, Pedroni E, Coray A, Jermann M, Rutz HP, Goitein G. Spot-scanning proton therapy for malignant soft tissue tumors in childhood: First experiences at the Paul Scherrer Institute. Int J Radiat Oncol Biol Phys. 2007 Feb 1;67(2):497-504. doi: 10.1016/j.ijrobp.2006.08.053. Epub 2006 Nov 2. PMID 17084557
- [Background] Weber DC, Rutz HP, Bolsi A, Pedroni E, Coray A, Jermann M, Lomax AJ, Hug EB, Goitein G. Spot scanning proton therapy in the curative treatment of adult patients with sarcoma: the Paul Scherrer institute experience. Int J Radiat Oncol Biol Phys. 2007 Nov 1;69(3):865-71. doi: 10.1016/j.ijrobp.2007.04.034. Epub 2007 Jul 2. PMID 17606333
- [Background] DeLaney TF, Trofimov AV, Engelsman M, Suit HD. Advanced-technology radiation therapy in the management of bone and soft tissue sarcomas. Cancer Control. 2005 Jan-Feb;12(1):27-35. doi: 10.1177/107327480501200104. PMID 15668650
- [Background] Brada M, Pijls-Johannesma M, De Ruysscher D. Proton therapy in clinical practice: current clinical evidence. J Clin Oncol. 2007 Mar 10;25(8):965-70. doi: 10.1200/JCO.2006.10.0131. No abstract available. PMID 17350945
- [Background] Bjork-Eriksson T, Bjelkengren G, Glimelius B. The potentials of proton beam radiation therapy in malignant lymphoma, thymoma and sarcoma. Acta Oncol. 2005;44(8):913-7. doi: 10.1080/02841860500355983. PMID 16332601
- [Background] Borden EC, Baker LH, Bell RS, Bramwell V, Demetri GD, Eisenberg BL, Fletcher CD, Fletcher JA, Ladanyi M, Meltzer P, O'Sullivan B, Parkinson DR, Pisters PW, Saxman S, Singer S, Sundaram M, van Oosterom AT, Verweij J, Waalen J, Weiss SW, Brennan MF. Soft tissue sarcomas of adults: state of the translational science. Clin Cancer Res. 2003 Jun;9(6):1941-56. PMID 12796356
- [Background] Tuma RS. Sometimes size doesn't matter: reevaluating RECIST and tumor response rate endpoints. J Natl Cancer Inst. 2006 Sep 20;98(18):1272-4. doi: 10.1093/jnci/djj403. No abstract available. PMID 16985244
- [Background] Zagars GK, Ballo MT, Pisters PW, Pollock RE, Patel SR, Benjamin RS. Preoperative vs. postoperative radiation therapy for soft tissue sarcoma: a retrospective comparative evaluation of disease outcome. Int J Radiat Oncol Biol Phys. 2003 Jun 1;56(2):482-8. doi: 10.1016/s0360-3016(02)04510-8. PMID 12738324
- [Background] Baur A, Reiser MF. Diffusion-weighted imaging of the musculoskeletal system in humans. Skeletal Radiol. 2000 Oct;29(10):555-62. doi: 10.1007/s002560000243. PMID 11127677
- [Background] Chenevert TL, Stegman LD, Taylor JM, Robertson PL, Greenberg HS, Rehemtulla A, Ross BD. Diffusion magnetic resonance imaging: an early surrogate marker of therapeutic efficacy in brain tumors. J Natl Cancer Inst. 2000 Dec 20;92(24):2029-36. doi: 10.1093/jnci/92.24.2029. PMID 11121466
- [Background] Hosseinzadeh K, Schwarz SD. Endorectal diffusion-weighted imaging in prostate cancer to differentiate malignant and benign peripheral zone tissue. J Magn Reson Imaging. 2004 Oct;20(4):654-61. doi: 10.1002/jmri.20159. PMID 15390142
- [Background] Namimoto T, Yamashita Y, Sumi S, Tang Y, Takahashi M. Focal liver masses: characterization with diffusion-weighted echo-planar MR imaging. Radiology. 1997 Sep;204(3):739-44. doi: 10.1148/radiology.204.3.9280252.
- [Background] Low RN, Gurney J. Diffusion-weighted MRI (DWI) in the oncology patient: value of breathhold DWI compared to unenhanced and gadolinium-enhanced MRI. J Magn Reson Imaging. 2007 Apr;25(4):848-58. doi: 10.1002/jmri.20864. PMID 17335018
- [Background] Hamstra DA, Rehemtulla A, Ross BD. Diffusion magnetic resonance imaging: a biomarker for treatment response in oncology. J Clin Oncol. 2007 Sep 10;25(26):4104-9. doi: 10.1200/JCO.2007.11.9610. PMID 17827460
- [Background] Einarsdottir H, Karlsson M, Wejde J, Bauer HC. Diffusion-weighted MRI of soft tissue tumours. Eur Radiol. 2004 Jun;14(6):959-63. doi: 10.1007/s00330-004-2237-0. Epub 2004 Feb 6. PMID 14767604
- [Background] Roberts C, Issa B, Stone A, Jackson A, Waterton JC, Parker GJ. Comparative study into the robustness of compartmental modeling and model-free analysis in DCE-MRI studies. J Magn Reson Imaging. 2006 Apr;23(4):554-63. doi: 10.1002/jmri.20529. PMID 16506143
- [Background] Jackson A, O'Connor JP, Parker GJ, Jayson GC. Imaging tumor vascular heterogeneity and angiogenesis using dynamic contrast-enhanced magnetic resonance imaging. Clin Cancer Res. 2007 Jun 15;13(12):3449-59. doi: 10.1158/1078-0432.CCR-07-0238. PMID 17575207
- [Background] Flickinger FW, Allison JD, Sherry RM, Wright JC. Differentiation of benign from malignant breast masses by time-intensity evaluation of contrast enhanced MRI. Magn Reson Imaging. 1993;11(5):617-20. doi: 10.1016/0730-725x(93)90002-u. PMID 8345775
- [Background] Knopp MV, Weiss E, Sinn HP, Mattern J, Junkermann H, Radeleff J, Magener A, Brix G, Delorme S, Zuna I, van Kaick G. Pathophysiologic basis of contrast enhancement in breast tumors. J Magn Reson Imaging. 1999 Sep;10(3):260-6. doi: 10.1002/(sici)1522-2586(199909)10:33.0.co;2-7. PMID 10508285
- [Background] Cella DF, Tulsky DS, Gray G, Sarafian B, Linn E, Bonomi A, Silberman M, Yellen SB, Winicour P, Brannon J, et al. The Functional Assessment of Cancer Therapy scale: development and validation of the general measure. J Clin Oncol. 1993 Mar;11(3):570-9. doi: 10.1200/JCO.1993.11.3.570. PMID 8445433
- [Background] Sugarbaker PH, Barofsky I, Rosenberg SA, Gianola FJ. Quality of life assessment of patients in extremity sarcoma clinical trials. Surgery. 1982 Jan;91(1):17-23. PMID 7054901
- [Background] Wang D, Kirsch DG, Okuno SH, Eisenberg BL, Kane JM, Li XA, Lucas D, Kraybill W, Chamberlain Wilmoth M RTOG 0630, A phase II trial of image guided preoperative radiotherapy for primary soft tissue sarcomas of the extremity. 2008.
- [Background] Zahlten-Hinguranage A, Bernd L, Ewerbeck V, Sabo D. Equal quality of life after limb-sparing or ablative surgery for lower extremity sarcomas. Br J Cancer. 2004 Sep 13;91(6):1012-4. doi: 10.1038/sj.bjc.6602104. PMID 15292924
- [Background] Onal C, Ozyar E. In regards to Sze et al.: Primary tumor volume of nasopharyngeal carcinoma: prognostic significance for local control (Int J Radiat Oncol Biol Phys 2004;59:21-27). Int J Radiat Oncol Biol Phys. 2005 Feb 1;61(2):629; author reply 629. doi: 10.1016/j.ijrobp.2004.10.006. No abstract available. PMID 15667986
- [Background] Davis AM, Wright JG, Williams JI, Bombardier C, Griffin A, Bell RS. Development of a measure of physical function for patients with bone and soft tissue sarcoma. Qual Life Res. 1996 Oct;5(5):508-16. doi: 10.1007/BF00540024. PMID 8973131
- [Background] Hua C, Gray JM, Merchant TE, Kun LE, Krasin MJ. Treatment planning and delivery of external beam radiotherapy for pediatric sarcoma: the St. Jude Children's Research Hospital experience. Int J Radiat Oncol Biol Phys. 2008 Apr 1;70(5):1598-606. doi: 10.1016/j.ijrobp.2007.12.013. Epub 2008 Jan 30. PMID 18234441
- [Background] Jastak Associates. Manual for the Wide Range Achievement Test - 3. Wilmington DE: Wide Range; 1993.
- [Background] Schreiber D, Bell RS, Wunder JS, O'Sullivan B, Turcotte R, Masri BA, Davis AM. Evaluating function and health related quality of life in patients treated for extremity soft tissue sarcoma. Qual Life Res. 2006 Nov;15(9):1439-46. doi: 10.1007/s11136-006-0001-4. Epub 2006 May 27. PMID 16732468
- [Background] Hanley MA, Jensen MP, Ehde DM, Hoffman AJ, Patterson DR, Robinson LR. Psychosocial predictors of long-term adjustment to lower-limb amputation and phantom limb pain. Disabil Rehabil. 2004 Jul 22-Aug 5;26(14-15):882-93. doi: 10.1080/09638280410001708896. PMID 15497917